CLINICAL TRIAL: NCT05673863
Title: The Efficacy of the Psychological Resilience Program for the Adolescent Girls Who Are Victims of Sexual Abuse
Brief Title: Resilience in Girls Victims of Sexual Abuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, GÜLGÜNDURAT, associate professor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SU-OKSAL-001
Record Dates: First submitted 2022-12-16; First posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-12

CONDITIONS: Child Sexual Abuse

STUDY DESIGN:
Intervention Model Description: The sample consisted of girls who agreed to participate in the study and one of their family members (mother, father, aunt, etc.).
Who Masked: Participant, Investigator
Masking Description: Children who met the criteria of the study and agreed to be included in the study were first divided according to age groups (11-13 years and 14-16 years) by block randomization and the sample group was formed. These individuals were then randomly assigned to the intervention and control groups by double-blinding method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychological resilience training program (Experimental): Children in the intervention group participated in a psychological resilience program organized as a group activity.
  Interventions: Behavioral: Psychological Resilience Program
- control group (No Intervention): Children in the control group did not receive any intervention. There was also no intervention for the family members accompanying the children.

INTERVENTIONS:
Behavioral: Psychological Resilience Program — The psychological resilience program was applied to the children in the intervention group twice a week for a total of 5 weeks. Each session consisted of 90 minutes of structured practice. The application is carried out using narrative therapy, cognitive behavioral therapy, psychodrama and analogy techniques, self-assessment and didactic teaching techniques. In addition, participants were engaged in self-regulation exercises and positive imagery activities. Each session includes practices on empathy, stress management, resilience, realistic and unrealistic thinking, optimism and pessimism, autonomy and humor related to resilience.
  Arms: Psychological resilience training program

SUMMARY:
İn this study, it was aimed to examine the effectiveness of the psychological resilience program for adolescent girls after sexual abuse.This study is a randomized controlled trial.

DETAILED DESCRIPTION:
Sexual abuse, which is a universal problem, affects the functioning of many institutions of society and can lead to lifelong physical, mental and social problems and health problems for children.The process of coping and adapting to stressful challenges such as sexual abuse is explained by psychological resilience.

Social support provided by parents, peers and professionals from the onset of sexual abuse contributes positively to children's lives and facilitates adaptation.Group therapies to be applied to abuse victims can increase perceived social support by reducing negative effects such as shame and stigmatization.

ELIGIBILITY:
Inclusion Criteria:

* Having applied to a child advocacy center due to sexual abuse
* Being a girl in the 11-18 age group
* The cognitive competence required to maintain the measurement tools and the training process to have
* Volunteering to participate in the research
* Being open to communication and cooperation
* No severe psychiatric disorder (such as psychosis, neurosis)
* The child can become literate (to be able to use assessment tools)

Exclusion Criteria:

* Not wanting to participate in the research
* To continue the group training or to fill in the measurement tools to be applied cognitive and physical dysfunction that would constitute an obstacle.

Ages: 11 Years to 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — participants were adolescent girls
Enrollment: 38 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
For children Resiliency Attitudes and Skills Profile (RASP) | 6 months
  The increase in the score obtained from the scale is associated with an increase in resilience. The aim is to define four sub-factors related to psychological resilience: (1) relationships and values, (2) insight and creativity, (3) independence and entrepreneurship, and (4) humor. The scale consists of 34 items on a 4-point Likert scale ranging from strongly disagree (1) to strongly agree (4)
For children Strengths and Difficulties Questionnaire (SDQ) Adolescent Form: | 6 months
  It consists of 24 items and is a 7-point Likert scale ranging from (7) Strongly agree to (1) Strongly disagree. The lowest score obtained from the scale is 24, and the highest score is 168. A high score indicates a high level of self-recovery power.
For children Resilience Scale(RS) | 6 months
  It consists of 24 items and is a 7-point Likert scale ranging from (7) Strongly agree to (1) Strongly disagree. The lowest score obtained from the scale is 24, and the highest score is 168. A high score indicates a high level of self-recovery power.

SECONDARY OUTCOMES:
For parents(Strengths and Difficulties Questionnaire Parent Form (SDQ) | 6 months
  The scale consists of 25 questions and five sub-dimensions, as in the child form. The sub-dimensions, attention deficit and hyperactivity, behavioral problems, emotional problems, and peer problems, show the difficulties experienced separately. The total difficulty score can be calculated by summing these four sub-dimensions. The social behaviors sub-dimension refers to strength.

OTHER OUTCOMES:
For parents Beck Depression Inventory (BDI): | 6 months
  The 21-item scale, each consisting of four options, includes assessments of how people have felt in the last week. A high score determines the severity of depressive symptoms.
For parents Beck Anxiety Scale (BAS) | 6 months
  The scale consists of 21 items and is a 4-point Likert-type self-assessment scale scored between 0 and 3. The questions aimed to evaluate how people have felt in the last week. The increase in the obtained score determines the high level of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: GÜLGÜN DURAT, PhD, Principal Investigator — Sakarya University
Locations (1):
- Sakarya University, Sakarya, Serdivan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No